CLINICAL TRIAL: NCT01673087
Title: Stress Biomarkers:Attaching Biological Meaning to Field Friendly Salivary Measures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James Abelson, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01MH093486-01A1 (NIH)
Record Dates: First submitted 2012-08-16; First posted 2012-08-27 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Stress
Keywords: stress biology; cortisol; adrenocorticotropin; salivary biomarkers
MeSH Terms: interventions — Metyrapone; Dexamethasone; Calcium Dobesilate; Cosyntropin; corticorelin ovine; Corticotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- laboratory HPA probes (Experimental): All subjects will be studied with multiple probes of HPA axis function over the course of one to two months:
  Metyrapone, oral, 750 mg, administered twice 3.5 hrs apart; Dexamethasone, oral, 1.5 mg administered once; oral, 0.25 mg administered once; Corticorelin ovine triflutate (CRH), intravenous, 100 mcg, administered once over 30 seconds; Cortrosyn (ACTH), intravenous, 250 mcg, administered once by bolus.
  Interventions: Drug: Metyrapone; Drug: Dexamethasone; Drug: Cortrosyn; Drug: Corticorelin ovine triflutate

INTERVENTIONS:
Drug: Metyrapone — 750 mcg, oral, administered twice, 3.5 hours apart
  Other Names: Metopirone
Drug: Dexamethasone — Administered twice:
  1.5 mg, oral, at 11 pm And 0.25 mg, oral, at bedtime at least one week before or after other administration.
  Other Names: Decadron
Drug: Cortrosyn — 250 mcg, IV, bolus, in the afternoon.
  Other Names: Cosyntropin
Drug: Corticorelin ovine triflutate — 100 mcg, IV, over 30 seconds, in the afternoon.
  Other Names: Acthrel; Corticotropin-Releasing Hormone

SUMMARY:
Cortisol is a stress hormone that can be measured in saliva. This has provided a convenient way to evaluate the biological impact of day-to-day stressors that people encounter as they go about their lives, since saliva is so easy to collect. However, the biological meaning of saliva cortisol measures has never been carefully examined. The goal of this study is to collect saliva from a large group of people as they go about their every-day lives, to measure their cortisol levels, and then study them in the laboratory where Investigators can learn more about how their stress response system (which produces cortisol) is really functioning. Investigators can then determine much more precisely what saliva cortisol levels really mean in terms of stress system biology. This will allow investigators to obtain much more useful information from the next decade of research on naturalistic stress and its biological impact using saliva cortisol measures, helping investigators to understand how stress undermines health and how to combat this effect.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy volunteers, ages 18 to 50 years

Exclusion Criteria:

* Pregnancy
* Irregular menses, medications or drugs that effect HPA axis
* Most psychiatric disorders
* Medical problems that effect HPA axis or increase risks involved in participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2012-10; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
cortisol levels | Primarily measuring change from pre-drug baseline to peak occuring about 20 minutes to an hour later
  cortisol measured in saliva and in blood.

SECONDARY OUTCOMES:
corticotropin (ACTH) | Primarily measuring change from pre-drug baseline to peak occuring about 10 minutes to an hour later
  ACTH will be measured in blood using chemoluminescence detection.

CONTACTS AND LOCATIONS:
Overall Officials: James L Abelson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States